CLINICAL TRIAL: NCT00681291
Title: Prospective, Randomized, Controlled, Third-Party Blinded Multicenter Evaluation of Strattice/LTM in the Repair of Inguinal Hernias
Brief Title: Strattice in Repair of Inguinal Hernias
Acronym: RING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LFC2007.04.01
Record Dates: First submitted 2008-05-15; First posted 2008-05-21 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-04

CONDITIONS: Hernia, Inguinal
Keywords: surgical mesh; inguinal hernia repair; chronic groin pain
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): lightweight polypropylene mesh
  Interventions: Device: Inguinal hernia repair with Ultrapro
- 2 (Active Comparator): Strattice
  Interventions: Device: Inguinal hernia repair with Strattice

INTERVENTIONS:
Device: Inguinal hernia repair with Ultrapro — surgical mesh (15x15cm) to support Lichtenstein repair
  Other Names: Ultrapro (Ethicon, Somerville NJ)
  Arms: 1
Device: Inguinal hernia repair with Strattice — Surgical mesh (10x16) used to support Lichtenstein repair
  Other Names: Strattice Reconstructive Tissue Matrix
  Arms: 2

SUMMARY:
This is a prospective, randomized, controlled, third-party blinded, multicenter, interventional evaluation of inguinal hernia repair comparing Strattice to light weight polypropylene mesh. Performance and outcomes measures to be compared include postoperative resumption of activities of daily living, nature and incidence of short- and long-term pain and complications, and incidence of hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* adult male
* symptomatic and palpable inguinal hernia
* open, elective, primary unilateral inguinal hernia repair

Exclusion Criteria:

* bilateral inguinal hernia repair
* BMI >35
* chronic immunosuppression, active chemo/radiation therapy, uncontrolled diabetes, severe liver disease or COPD
* chronic prostatitis, orchitis, testicular pain
* local or systemic infection at time of repair
* known collagen disorder
* chronic pain syndrome or under active pain management

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bellows, MD, FACS, Principal Investigator — Tulane University; Samir Awad, MD, FACS, Principal Investigator — Baylor College of Medicine; Robert Fitzgibbons, MD, FACS, Principal Investigator — Creighton University
Locations (8):
- United States (8):
  - Hospital of St Raphael, New Haven, Connecticut
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Creighton University, Omaha, Nebraska
  - Regional Surgical Associates, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

REFERENCES:
- [Derived] Bellows CF, Shadduck PP, Helton WS, Fitzgibbons RJ. The design of an industry-sponsored randomized controlled trial to compare synthetic mesh versus biologic mesh for inguinal hernia repair. Hernia. 2011 Jun;15(3):325-32. doi: 10.1007/s10029-010-0773-x. Epub 2011 Jan 8. PMID 21222008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on April 11, 2008 and last subject was enrolled on February 12, 2010.
Groups:
- 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r: lightweight polypropylene mesh
- 2Strattice (Utilized for Inguinal Hernia Repair): Strattice
Period: Overall Study
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Started | 88 | 84
Completed | 75 | 57
Not Completed | 13 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair) | Total
Number analyzed (Participants) | 88 | 84 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.78) | 55.2 (14.53) | 55.8 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 88 | 84 | 172
Region of Enrollment [Number; unit: participants]
  United States | 88 | 84 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Activities Assessment Scale at 3 Months
Description: The AAS includes 13 items covering a broad sample of sedentary, movement-related and graded-intensity physical activities. Respondents are asked to rate the degree of difficulty performing each of these activities in the previous 24 hours on a 5-point scale from "No difficulty = 1" to "Not able to do it = 5." The AAS has three subscales: sedentary activities (items 1-4); ambulatory activities (items 6-8); work/exercise activities (items 11-13). The AAS total and subscale scores are transformed to produce a range of 0-100, with higher values indicating greater functional activity. Subjects completed the assessment at baseline, 3 months, 6 months, 12 months and 24 months. It is the change from baseline to 3, 6, 12 and 24 months which is the primary outcome measure (Baseline calculated value minus time point calculated value). Therefore, a negative number indicates an increase in activity from baseline.
Time Frame: Baseline to 3 Months
Population: Of the 88 participants in Arm 1 who started the study, 81 completed the Activities Assessment Scale at 3 months. Of the 84 participants in Arm 2 who started the study, 77 completed the Activities Assessment Scale at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Number analyzed (Participants) | 81 | 77
units on a scale | -7.49 (8.961) | -6.12 (8.666)

2. Primary Outcome: Change From Baseline in Activities Assessment Scale at 6 Months
Description: The AAS includes 13 items covering a broad sample of sedentary, movement-related and graded-intensity physical activities. Respondents are asked to rate the degree of difficulty performing each of these activities in the previous 24 hours on a 5-point scale from "No difficulty" to "Not able to do it." The AAS has three subscales: sedentary activities (items 1-4); ambulatory activities (items 6-8); work/exercise activities (items 11-13). The AAS total and subscale scores are transformed to produce a range of 0-100, with higher values indicating greater functional activity. Subjects completed the assessment at baseline, 3 months, 6 months, 12 months and 24 months. It is the change from baseline to 3, 6, 12 and 24 months which is the primary outcome measure (Baseline calculated value minus time point calculated value). Therefore, a negative number indicates an increase in activity from baseline.
Time Frame: Baseline to 6 Months
Population: Of the 88 participants in Arm 1 who started the study, 83 completed the Activities Assessment Scale at 6 months. Of the 84 participants in Arm 2 who started the study, 70 completed the Activities Assessment Scale at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Number analyzed (Participants) | 83 | 70
units on a scale | -8.17 (9.475) | -7.20 (8.818)

3. Primary Outcome: Change From Baseline in Activities Assessment Scale at 12 Months
Description: as for outcome 2
Time Frame: Baseline to 12 Months
Population: Of the 88 participants in Arm 1 who started the study, 83 completed the Activities Assessment Scale at 12 months. Of the 84 participants in Arm 2 who started the study, 70 completed the Activities Assessment Scale at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Number analyzed (Participants) | 83 | 70
units on a scale | -8.78 (9.221) | -7.61 (9.059)

4. Primary Outcome: Change From Baseline in Activities Assessment Scale at 24 Months
Description: as for outcome 2
Time Frame: Baseline to 24 Months
Population: Of the 88 participants in Arm 1 who started the study, 75 completed the Activities Assessment Scale at 24 months. Of the 84 participants in Arm 2 who started the study, 57 completed the Activities Assessment Scale at 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Number analyzed (Participants) | 75 | 57
units on a scale | -7.57 (8.098) | -7.53 (9.356)

ADVERSE EVENTS:
Arm/Group | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r | 2Strattice (Utilized for Inguinal Hernia Repair)
Serious Adverse Events (participants affected / at risk) | 2/88 | 4/84
Other Adverse Events (participants affected / at risk) | 47/88 | 49/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r (N=88) | 2Strattice (Utilized for Inguinal Hernia Repair) (N=84)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1lightweight Polypropylene Mesh(Utilized for Inguinal Hernia r (N=88) | 2Strattice (Utilized for Inguinal Hernia Repair) (N=84)
Inguinal Hernia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Local Swelling (General disorders) | 5 (5) | 2 (2)
Incision Site Pain (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
C-Reactive Protein Increased (Investigations) | 15 (15) | 21 (21)
Groin Pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 4 (4)
Hypoaethesia (Nervous system disorders) | 2 (2) | 8 (8)
Testicular Pain (Reproductive system and breast disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should Institution/PI/coPI/other staff want to publish information, data, or orally communicate,a complete copy of information/data will be provided to the Sponsor for review and comment at least 30 days prior to 1st submission. If Sponsor determines proposed publication/oral communication contains patentable or proprietary subject matter (requiring protection),Institution will delay for at least 90 days following the Sponsor's receipt of such copy for the purpose of filing patent applications.